CLINICAL TRIAL: NCT06989762
Title: Use of an Intraabdominal Pressure Monitoring Urinary Catheter After Cardiac Surgery to Improve Kidney Perfusion Pressure: A Randomized Controlled Trial
Brief Title: Intraabdominal Pressure Monitoring Urinary Catheter and Kidney Perfusion Pressure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dang Tan Phat (Other)
Responsible Party: Sponsor-Investigator, Dang Tan Phat, Assistant Clinical Professor, Department of Anesthesiology & Perioperative Care, University of California, Irvine, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2756
Record Dates: First submitted 2025-04-15; First posted 2025-05-25 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Intra-Abdominal Pressure; Renal Perfusion Pressure; Cardiac Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group - Standard ICU Care with Conventional Foley (Active Comparator): Participants will receive standard ICU care after cardiac surgery with a conventional Foley catheter. Blood pressure management will follow routine ICU protocols without intra-abdominal pressure (IAP) monitoring.
  Interventions: Device: Conventional Foley Catheter(Medline)
- Intervention Group - IAP Monitoring and Renal Perfusion Pressure Optimization (Experimental): Participants will receive standard ICU care after cardiac surgery with an IAP-monitoring Foley catheter. Blood pressure will be adjusted based on IAP readings to optimize renal perfusion pressure(41mmHg).
  Interventions: Device: Accuryn Foley Catheter

INTERVENTIONS:
Device: Conventional Foley Catheter(Medline) — The Conventional Foley Catheter is a standard urinary catheter used in ICU care to monitor urine output. It does not have intra-abdominal pressure (IAP) monitoring capabilities.
  Arms: Control Group - Standard ICU Care with Conventional Foley
Device: Accuryn Foley Catheter — The Accuryn Foley Catheter is an FDA-approved urinary catheter with continuous intra-abdominal pressure (IAP) monitoring capability.
  Arms: Intervention Group - IAP Monitoring and Renal Perfusion Pressure Optimization

SUMMARY:
The goal of this clinical trial is to determine whether monitoring intra-abdominal pressure (IAP) and adjusting blood pressure accordingly to maintain optimal renal perfusion pressure can reduce the risk of acute kidney injury (AKI) after cardiac surgery.

The main question this study aims to answer is:

- Does IAP-guided blood pressure management improve renal perfusion and lower AKI rates in cardiac surgery patients?

Participants will be randomly assigned to one of two groups:

* Control Group: Standard ICU care with a conventional Foley catheter.
* Intervention Group: Standard ICU care with an IAP-monitoring Foley catheter, where blood pressure is adjusted based on IAP readings to optimize renal perfusion pressure.

All participants will undergo routine blood and urine tests to assess kidney function during their hospital stay.

This study will help determine whether IAP-based hemodynamic management can improve postoperative kidney outcomes and provide a new strategy for AKI prevention in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults Undergoing cardiac surgery with cardiopulmonary bypass
* Left ventricular ejection fraction (LVEF) < 50%

Exclusion Criteria:

* Current pregnancy
* ESRD or AKI on dialysis
* Currently on ECMO or Impella
* Emergent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Acute Kidney Injury (AKI) as defined by KDIGO Criteria | Perioperative.
  Acute Kidney Injury will be defined using the KDIGO criteria: an increase in serum creatinine by ≥0.3 mg/dL within 48 hours or an increase to ≥1.5 times the baseline.

SECONDARY OUTCOMES:
ICU Length of Stay | Perioperative
  The number of days from the day of surgery until discharge from the ICU
Hospital Length of Stay | Perioperative
  The number of days from the day of surgery until discharge from the hospital (including both ICU and general ward)

CONTACTS AND LOCATIONS:
Locations (1):
- UCI Medical Center, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No
The IPB will be kept for this study only. Will not share with any other study

REFERENCES:
- [Background] Chen SS, Chen WC, Hayakawa S, Li PC, Chien CT. Acute urinary bladder distension triggers ICAM-1-mediated renal oxidative injury via the norepinephrine-renin-angiotensin II system in rats. J Formos Med Assoc. 2009 Aug;108(8):627-35. doi: 10.1016/s0929-6646(09)60383-1. PMID 19666350
- [Background] Hertzberg D, Sartipy U, Lund LH, Ryden L, Pickering JW, Holzmann MJ. Heart failure and the risk of acute kidney injury in relation to ejection fraction in patients undergoing coronary artery bypass grafting. Int J Cardiol. 2019 Jan 1;274:66-70. doi: 10.1016/j.ijcard.2018.09.092. Epub 2018 Sep 28. PMID 30297189
- [Background] Gao Y, Wang C, Li J, Ji B, Wang J, Yan F, Wang Y. Mild and moderate to severe early acute kidney injury following cardiac surgery among patients with heart failure and preserved vs. mid-range vs. reduced ejection fraction: A retrospective cohort study. Eur J Anaesthesiol. 2022 Aug 1;39(8):673-684. doi: 10.1097/EJA.0000000000001713. Epub 2022 Jul 5. PMID 35791895
- [Background] Kopitko C, Medve L, Gondos T. The value of combined hemodynamic, respiratory and intra-abdominal pressure monitoring in predicting acute kidney injury after major intraabdominal surgeries. Ren Fail. 2019 Nov;41(1):150-158. doi: 10.1080/0886022X.2019.1587467. PMID 30909772
- [Background] Dalfino L, Sicolo A, Paparella D, Mongelli M, Rubino G, Brienza N. Intra-abdominal hypertension in cardiac surgery. Interact Cardiovasc Thorac Surg. 2013 Oct;17(4):644-51. doi: 10.1093/icvts/ivt272. Epub 2013 Jul 2. PMID 23820668
- [Background] Sun J, Sun H, Sun Z, Yang X, Zhou S, Wei J. Intra-abdominal hypertension and increased acute kidney injury risk: a systematic review and meta-analysis. J Int Med Res. 2021 May;49(5):3000605211016627. doi: 10.1177/03000605211016627. PMID 34053324
- [Background] Hobson CE, Yavas S, Segal MS, Schold JD, Tribble CG, Layon AJ, Bihorac A. Acute kidney injury is associated with increased long-term mortality after cardiothoracic surgery. Circulation. 2009 May 12;119(18):2444-53. doi: 10.1161/CIRCULATIONAHA.108.800011. Epub 2009 Apr 27. PMID 19398670
- [Background] Engelman DT, Schwann TA. Commentary: A little is way too much: What we have learned about perioperative acute kidney injury. J Thorac Cardiovasc Surg. 2021 Jul;162(1):153-154. doi: 10.1016/j.jtcvs.2019.12.100. Epub 2020 Jan 21. No abstract available. PMID 32061391
- [Background] Priyanka P, Zarbock A, Izawa J, Gleason TG, Renfurm RW, Kellum JA. The impact of acute kidney injury by serum creatinine or urine output criteria on major adverse kidney events in cardiac surgery patients. J Thorac Cardiovasc Surg. 2021 Jul;162(1):143-151.e7. doi: 10.1016/j.jtcvs.2019.11.137. Epub 2020 Jan 9. PMID 32033818
- [Background] Dang PT, Lopez BE, Togashi K. A Decrease in Effective Renal Perfusion Pressure Is Associated With Increased Acute Kidney Injury in Patients Undergoing Cardiac Surgery. Cureus. 2023 Sep 11;15(9):e45036. doi: 10.7759/cureus.45036. eCollection 2023 Sep. PMID 37829983